CLINICAL TRIAL: NCT01743456
Title: Effect of Depth of Anaesthesia on Postoperative Cognitive Decline in Patients Undergoing Coronary Artery Bypass Graft Surgery - a Prospectively Randomized Controlled Study
Brief Title: Depth of Anaesthesia and Postoperative Cognitive Decline in Patients Undergoing Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KHC11-001
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2013-01

CONDITIONS: Cardiac Bypass Surgery in Adult Patients 65 Years and Older; Postoperative Cognitive Dysfunction; Postoperative Delirium
Keywords: Postoperative cognitive dysfunction; Coronary artery bypass graft surgery; Postoperative cognitive improvement; Postoperative delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Current practice (BIS and rSO2 blinded) (No Intervention)
- Targeted intra-operative depth of anaesthesia (Experimental)
  Interventions: Other: Targeted intra-operative depth of anaesthesia

INTERVENTIONS:
Other: Targeted intra-operative depth of anaesthesia — The intervention group receives isoflurane at a concentration that results in a BIS value between 40-60 intra-operatively.
  Arms: Targeted intra-operative depth of anaesthesia

SUMMARY:
Post-Operative Cognitive Decline (POCD) is common after cardiac surgery and associated with increased morbidity and mortality. The pathophysiology of POCD is only poorly understood. Causes include hypoperfusion, microemboli and the systemic inflammatory response, which result in a reduction of cerebral oxygen delivery.

Cerebral oxygenation can be monitored non-invasively by measuring frontal lobe oxygen saturation (rSO2).

The bispectral index (BIS) of the electroencephalogram is widely known to measure depth of anaesthesia, and there is a high correlation between BIS, a dimensionless calculated number between 0 and 100, and clinical criteria of sedation. With BIS below 60 recall is extremely low.

The investigators demonstrated recently that inappropriately high levels of anaesthesia may be associated with poorer long-term outcomes in cognition after non-cardiac surgery (Ballard et al. 2012). Whether optimisation of the depth of anaesthesia and cerebral oxygenation has an effect on postoperative cognitive function in patients undergoing cardiac surgery is unknown.

The investigators hypothesize that the incidence of POCD in elderly patients (> 65 years old) at 6 weeks is less with mildly deep anaesthesia (BIS 50 +- 10) and optimised rSO2 (interventions when rSO2 drops below 15% of baseline reading) when compared with current practice (BIS blinded anaesthesia, reflecting moderately to highly deep anaesthesia and blinded rSO2 measurements).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective coronary artery bypass graft surgery
* patients at 65 years of age and older

Exclusion Criteria:

* diseases of the central nervous system including dementia
* inadequate knowledge of English
* a current or past psychiatric illness
* current use of tranquilizers or antidepressants
* severe visual, auditory, or motor handicap

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive decline after bypass surgery | Six weeks after bypass surgery

SECONDARY OUTCOMES:
Incidence of postoperative cognitive decline 5 days and 1 year after bypass surgery | Five days and one year postoperatively
Difference in degree of postoperative cognitive decline at 5 days, 6 weeks or 1 year after bypass surgery | 5days, 6 weeks or 1 year postoperatively
Postoperative Delirium | 3-5 days postoperatively
Postoperative central nervous system and myocardial biochemical markers | up to 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: David Green, FRCA, MBA, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, Denmark Hill, United Kingdom

REFERENCES:
- [Background] Ballard C, Jones E, Gauge N, Aarsland D, Nilsen OB, Saxby BK, Lowery D, Corbett A, Wesnes K, Katsaiti E, Arden J, Amoako D, Prophet N, Purushothaman B, Green D. Optimised anaesthesia to reduce post operative cognitive decline (POCD) in older patients undergoing elective surgery, a randomised controlled trial. PLoS One. 2012;7(6):e37410. doi: 10.1371/journal.pone.0037410. Epub 2012 Jun 15. PMID 22719840